CLINICAL TRIAL: NCT01255111
Title: Adaptation to Nocturnal Noninvasive Ventilation in Patients With Chronic Respiratory Failure
Brief Title: Adaptation to Nocturnal Noninvasive Ventilation in Patients With Chronic Respiratory Failure (ROOMILA)
Acronym: ROOMILA
Status: Completed | Type: Observational
Sponsor: Groupe de Recherche sur le Handicap Respiratoire (Other)
Responsible Party: Pr. Antoine CUVELIER, GRHV - UPRES EA3830
Other Study IDs: 2010AC1
Record Dates: First submitted 2010-12-04; First posted 2010-12-07 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Respiratory Failure
Keywords: Chronic respiratory failure; Noninvasive ventilation; Patient-ventilator interactions; Sleep; Sleep fragmentation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
BACKGROUND: Adaptation to noninvasive ventilation (NIV) is a critical step for acceptability and efficacy of this treatment during sleep in patients with chronic respiratory failure.

AIM: To study the variability of patient-ventilator interactions during the first nights after initiation to NIV. Recorded data will be analyzed in part by dedicated tools from the non-linear dynamics theory.

PATIENTS AND METHODS: Patients with chronic respiratory failure at stable state and indicated to home NIV will be included. All patients will perform three polysomnographies (under spontaneous breathing at D1 and under NIV at D2 and D15 after NIV initiation). All ventilatory physiological data (pressure, flow, patient-ventilator interactions, oxygen saturation, non intentional leaks) will be recorded during sleep under NIV in the Sleep Laboratory of the Department and secondarily related to sleep architecture and quality of sleep.

EXPECTED RESULTS: This study will identify objective parameters that are associated to a satisfactory adaptation to nocturnal NIV.

ELIGIBILITY:
Inclusion Criteria:

* Chronic respiratory failure with indication to domiciliary NIV according to the international guidelines.

Exclusion Criteria:

* Decompensated respiratory failure attested by a pH <7.35,
* Modification of respiratory symptoms during the four previous weeks, including signs of broncho-pulmonary infection,
* Respiratory frequency >30/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic respiratory failure at stable state who are indicated to domiciliary noninvasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-10; Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Antoine CUVELIER, MD, PhD, Principal Investigator — Groupe de Recherche sur le Handicap Ventilatoire
Locations (1):
- Pulmonary & Respiratory Intensive Care Department - Rouen University Hospital, Rouen, France